CLINICAL TRIAL: NCT05139030
Title: A Phase 3, Randomized, Double-Blind, Multicenter, Active-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of EXPAREL Admixed With Bupivacaine Hydrochloric Acid (HCl) vs. Bupivacaine HCl Administered Via Adductor Canal Block for Postsurgical Analgesia in Subjects Undergoing Primary Unilateral Total Knee Arthroplasty
Brief Title: Phase 3 Adductor Canal Block With EXPAREL in Subjects Undergoing Primary Unilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-335
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis; Pain Management
Keywords: EXPAREL; bupivacaine; analgesic; Adductor Canal Block; TKA; knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only study drug administrators (anesthesiologists) will be unblinded to perform the block procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: EXPAREL admix arm (Experimental): subjects randomized to this treatment arm will receive 10 mL (133 mg) EXPAREL admixed with 10 mL (50 mg) 0.5% bupivacaine HCl
  Interventions: Drug: bupivacaine liposome injectable suspension
- Cohort 1: Bupivacaine HCl arm (Active Comparator): subjects randomized to this treatment arm will receive 10 mL (50 mg) 0.5% bupivacaine HCl mixed with 10 mL normal saline
  Interventions: Drug: Bupivacaine Hydrochloride
- Cohort 2: EXPAREL admix arm (Experimental): subjects randomized to this treatment arm will receive 10 mL (133 mg) EXPAREL admixed with 10 mL (50 mg) 0.5% bupivacaine HCl
  Interventions: Drug: bupivacaine liposome injectable suspension
- Cohort 2: Bupivacaine HCl arm (Active Comparator): subjects randomized to this treatment arm will receive 10 mL (50 mg) 0.5% bupivacaine HCl mixed with 10 mL normal saline
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: bupivacaine liposome injectable suspension — Adductor canal block with EXPAREL
  Other Names: EXPAREL
  Arms: Cohort 1: EXPAREL admix arm; Cohort 2: EXPAREL admix arm
Drug: Bupivacaine Hydrochloride — Adductor Canal Block with bupivacaine HCl
  Arms: Cohort 1: Bupivacaine HCl arm; Cohort 2: Bupivacaine HCl arm

SUMMARY:
The purpose of the study is to compare magnitude of postsurgical analgesic effect in different groups following a single dose of study drug when administered via adductor canal block in subjects undergoing primary unilateral total knee arthroplasty.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, active-controlled study in approximately 160 subjects undergoing primary unilateral TKA under spinal anesthesia. The study will have 2 cohorts, enrolling in parallel.

Cohort 1 -Pharmacokinetics (PK), pharmacodynamics (PD), Efficacy, and Safety, Cohort 2 -Efficacy and Safety

An adaptive study design will be used in this study. An interim analysis to evaluate the sample size assumptions and evaluate futility will occur when a total of approximately 80 subjects (40 subjects in each arm) combined from either Cohort 1 or Cohort 2 have enrolled and provided complete assessment data for the primary efficacy outcome.

The time from study drug administration until the end of participation is Post-operative day (POD) 14 (±3 days). Therefore, subjects may participate in the study for up to 62 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ages 18 or older at screening.
2. Indicated to undergo primary unilateral total knee arthroplasty under spinal anesthesia.
3. Primary indication for TKA is degenerative osteoarthritis of the knee.
4. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
5. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.
6. Body Mass Index (BMI) ≥18 and <40 kg/m2.

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine HCl, NSAIDs).
2. Planned concurrent surgical procedure (e.g., bilateral TKA).
3. Undergoing unicompartmental TKA or revision TKA.
4. Concurrent painful physical condition (e.g., arthritis, fibromyalgia, cancer) that may require analgesic treatment with NSAIDs or opioids in the post dosing period for pain that is not strictly related to the knee surgery and which, in the Investigator's opinion, may confound the post dosing assessments.
5. Inadequate sensory function below the knee as assessed by the Investigator.
6. History of contralateral TKA within 1 year.
7. Previous open knee surgery on the knee being considered for TKA. Prior arthroscopy is permitted.
8. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
9. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
10. Previous participation in an EXPAREL study.
11. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, could interfere with study assessments or compliance.
12. Currently pregnant, nursing, or planning to become pregnant during the study.
13. Clinically significant medical disease that, in the opinion of the Investigator, would make participation in a clinical study inappropriate. This includes diabetic neuropathy, coagulation or bleeding disorders, severe peripheral vascular disease, renal insufficiency, hepatic dysfunction, or other conditions that would constitute a contraindication to participation in the study.
14. Currently on a neuromodulating agent (e.g., gabapentin, pregabalin [Lyrica], duloxetine [Cymbalta], etc.)].
15. Current use of systemic glucocorticoids within 30 days of randomization in this study.
16. Use of dexmedetomidine HCl (Precedex®) or clonidine within 3 days of study drug administration.
17. Any use of marijuana [including Tetrahydrocannabinol (THC) and Cannabidiol (CBD)] within 30 days prior to randomization, or planned use during the course of the study.
18. Chronic opioid use (average ≥30 oral morphine equivalents/day) within 30 days prior to randomization.

Given the coronavirus disease 2019 (COVID-19) pandemic, if there is a concern about a subject's recent or potential exposure to COVID-19, or if the subject is not medically fit/cleared for surgery due to suspected COVID-19 illness/symptoms, the subject must be excluded per Exclusion criterion #13.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Nevins, Study Director — Pacira Pharmaceuticals, Inc
Locations (6):
- United States (6):
  - Woodland International Research Group, Little Rock, Arkansas
  - Lotus Clinical Research, Pasadena, California
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - HD Research- Legent Orthopedic Hospital, Carrollton, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gadsden J, Gonzales J, Saha P. Plain language summary of a pain medication (liposomal bupivacaine) for pain relief after knee replacement surgery. Pain Manag. 2025 Dec 19:1-10. doi: 10.1080/17581869.2025.2592701. Online ahead of print. PMID 41416686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 6 sites between January 2022 and July 2022. The first participant was enrolled on January 18, 2022 and the last participant was enrolled in June 08, 2022.
Pre-assignment Details: Of 340 screened participants, 167 met inclusion criteria and were randomized to treatment within Cohort 1 or Cohort 2. Overall results are presented per treatment arm including participants from both cohorts 1 + 2
Groups:
- Cohort 1 + 2: EXPAREL Admix Arm: subjects randomized to this treatment arm received 10 mL (133 mg) EXPAREL admixed with 10 mL (50 mg) 0.5% bupivacaine HCl
  bupivacaine liposome injectable suspension: Adductor canal block with EXPAREL
- Cohort 1 + 2: Bupivacaine HCl Arm: subjects randomized to this treatment arm received 10 mL (50 mg) 0.5% bupivacaine hydrochloric acid (HCl) mixed with 10 mL normal saline
  Bupivacaine Hydrochloride: Adductor Canal Block with bupivacaine HCl
Period: Overall Study
Arm/Group | Cohort 1 + 2: EXPAREL Admix Arm | Cohort 1 + 2: Bupivacaine HCl Arm
Started | 85 | 82
Completed | 84 | 77
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Failure to meet continuation criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of all participants for whom baseline characteristics were measured, in each cohort and in the entire study population (total)
Groups:
- Cohort 1 + 2: Bupivacaine HCl Arm: subjects randomized to this treatment arm received 10 mL (50 mg) 0.5% bupivacaine HCl mixed with 10 mL normal saline
  Bupivacaine Hydrochloride: Adductor Canal Block with bupivacaine HCl
- Total: Total of all reporting groups
Arm/Group | Cohort 1 + 2: EXPAREL Admix Arm | Cohort 1 + 2: Bupivacaine HCl Arm | Total
Number analyzed (Participants) | 85 | 81 | 166
Age, Categorical [Count of Participants; unit: Participants] — Population: Results presented are the combined participants of cohort 1 + cohort 2 treated with EXPAREL admixed with bupivacaiane HC1 and the combined participants of cohort 1 + cohort 2 treated with bupivacine HCI alone
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 54 | 53 | 107
    >=65 years | 31 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Results presented are the combined participants of cohort 1 + cohort 2 treated with EXPAREL admixed with bupivacaiane HC1 and the combined participants of cohort 1 + cohort 2 treated with bupivacine HCI alone
  years | 62.00 (7.049) | 62.21 (8.402) | 62.10 (7.716)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Results presented are the combined participants of cohort 1 + cohort 2 treated with EXPAREL admixed with bupivacaiane HC1 and the combined participants of cohort 1 + cohort 2 treated with bupivacine HCI alone
  Participants
    Female | 42 | 39 | 81
    Male | 43 | 42 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Measure Analysis Population Description: Results presented are the combined participants of cohort 1 + cohort 2 treated with EXPAREL admixed with bupivacaiane HC1 and the combined participants of cohort 1 + cohort 2 treated with bupivacine HCI alone
  Participants
    Hispanic or Latino | 21 | 12 | 33
    Not Hispanic or Latino | 64 | 66 | 130
    Unknown or Not Reported | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Results presented are the combined participants of cohort 1 + cohort 2 treated with EXPAREL admixed with bupivacaiane HC1 and the combined participants of cohort 1 + cohort 2 treated with bupivacine HCI alone
  Participants
    Race: White | 67 | 63 | 130
    Race: Black/African American | 14 | 15 | 29
    Race: Other | 4 | 3 | 7
Region of Enrollment [Number; unit: participants] — Population: Results presented are the combined participants of cohort 1 + cohort 2 treated with EXPAREL admixed with bupivacaiane HC1 and the combined participants of cohort 1 + cohort 2 treated with bupivacine HCI alone
  participants
    United States | 85 | 81 | 166
ASA classification [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical classification system is a grading system to determine the health of a person before a surgical procedure that requires anesthesia. The ASA classification was performed at baseline.
  ASA 1: a normal healthy patient ASA 2: a patient with mild systemic disease ASA 3: a patient with severe disease A lower ASA classification denotes better outcome
  Participants
    ASA 1 | 21 | 21 | 42
    ASA 2 | 62 | 56 | 118
    ASA 3 | 2 | 3 | 5
    Unknown | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kilograms/m^2] | 31.43 (4.786) | 32.74 (4.955) | 32.07 (4.899)
Body mass index, categorical [Count of Participants; unit: Participants]
  <25 kg/m^2 | 5 | 7 | 12
  25 to <30 kg/m^2 | 32 | 14 | 46
  >=30 kg/m^2 | 48 | 60 | 108
Worst pain intensity (NRS) [Mean (Standard Deviation); unit: units on a scale] — Worst pain intensity scores on a numeric rating scale ranging from 0 to 10,where 0 equals no pain and10 equals the worst possible pain, in the last 30 days of baseline. Mean score is provided The total range is 0 (no pain) to 10 (worst possible pain). Higher values on the scale represent worse outcome.
  units on a scale | 7.2 (2.03) | 7.4 (2.32) | 7.3 (2.17)
Average pain intensity (NRS) [Mean (Standard Deviation); unit: units on a scale] — Average pain intensity scores on a numeric rating scale ranging from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, in the last 30 days of baseline. Mean score is provided. The total range is 0 (no pain) to 10 (worst possible pain). Higher values on the scale represent worse outcome.
  units on a scale | 5.2 (2.32) | 5.3 (2.22) | 5.2 (2.27)

OUTCOME MEASURES:

1. Primary Outcome: NRS Scores Through 96 Hours Post-surgery
Description: The numeric rating scale pain intensity scores ranging from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, from 0 to 96 hours post-surgery. For each subject, the area under the curve was derived using the trapezoidal rule on the pain scores adjusted for opioid pain medication using the observed and imputed values. Area under the curve started with the first pain assessment obtained after surgery and use all subsequent pain assessments up to 96 hours post-surgery. Pain scores were taken at 5 interval point: 0 hours, 24 hours, 48 hours, 72 hours, and 96 hours. There were also unscheduled pain scores measured before opioid consumption also included in the area under the curve calculation. The area under the curve ranged from 0 to 960. Higher scores represent a worse outcome.
Time Frame: 0 to 96 hours post-surgery
Population: The analysis was performed on the efficacy analysis set which included all participants in the safety analysis set who underwent the planned surgery and had at least one post-drug administration NRS pain assessment. Results presented correspond to the combined population for cohorts 1 + 2 of each treatment arm
Measure: Mean (Standard Deviation); unit: units on a scale*hours
Groups:
- Cohort 1 + 2 EXPAREL ADMIX ARM: Subjects randomized to this treatment arm received 10 mL (133 mg) EXPAREL admixed with 10 mL (50 mg) 0.5% bupivacaine hydrochloric acid (HCI)
  Bupivacaine liposome injectable suspension Adductor canal block with EXPAREL
- Cohort 1 + 2 BUPIVACAINE HCI ARM: Subjects randomized to this treatment arm received 10 mL (50 mg) 0.5% bupivacaine HCI mixed with 10 mL normal saline Bupivacaine Hydrochloride Adductor Canal Block with bupivacaine HCI
Arm/Group | Cohort 1 + 2 EXPAREL ADMIX ARM | Cohort 1 + 2 BUPIVACAINE HCI ARM
Number analyzed (Participants) | 85 | 81
units on a scale*hours | 594.4 (191.65) | 650.1 (178.95)
Statistical Analysis 1: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; The superiority of EXPAREL admixed to bupivacaine HCI was evaluated using the Efficacy Analysis Set; Test type: Superiority — A one-sided hypothesis test was performed at alpha=0.025 level of significance comparing EXPAREL admix and bupivacaine HCI; p = 0.0074, ANCOVA; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Mean Difference (Final Values) = -65.8, 95% CI 2-sided [-118.7 to -12.9], Standard Error of Mean 26.97

2. Secondary Outcome: Postsurgical Opioid Consumption Through 96 Hours Post-surgery
Description: Total postsurgical opioid consumption in mg oral morphine equivalents (OMED) from 0 to 96 hours post-surgery.
Time Frame: 0 to 96 hours post-surgery
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams oral morphine equivalents
Groups:
- Cohort 1 + 2 EXPAREL ADMIX ARM: Subjects randomized to this treatment arm received 10 mL (133 mg) EXPAREL admixed with 10 mL (50 mg) 0.5% bupivacaine HCI
  Bupivacaine liposome injectable suspension Adductor canal block with EXPAREL
Arm/Group | Cohort 1 + 2 EXPAREL ADMIX ARM | Cohort 1 + 2 BUPIVACAINE HCI ARM
Number analyzed (Participants) | 85 | 81
milligrams oral morphine equivalents | 109.19 (54.420) | 136.91 (48.284)
Statistical Analysis 1: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; The superiority of EXPAREL admixed to bupivacaine HCI was evaluated using the Efficacy Analysis Set; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0018, ANCOVA; Total opioid consumption was transformed to log scale. Main effect of treatment, covariates: pooled Investigator site (categorical); age (continuous); Mean Ratio = 0.77, 95% CI 2-sided [0.64 to 0.92]

3. Secondary Outcome: Time to First Opioid
Description: Time to first opioid consumption post-surgery
Time Frame: 0 to 96 hours post-surgery
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Cohort 1 + 2 EXPAREL ADMIX ARM | Cohort 1 + 2 BUPIVACAINE HCI ARM
Number analyzed (Participants) | 85 | 81
hours | 4.15 [3.80 to 4.83] | 3.63 [2.98 to 4.05]
Statistical Analysis 1: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.0127, Cox proportional hazards model; Cox proportional hazard model: treatment as main effect, pooled Investigator site as categorical, and age and height as continuous covariates; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.51 to 0.96]

4. Secondary Outcome: NRS Scores
Description: Worst and average NRS pain intensity scores at 24h, 48h, 72h and 96h from the end of surgery Worst and average pain intensity scores on a numeric rating scale ranging from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, from 0 to 24 hours, 24 to 48 hours, 48 to 72 hours, and 72 to 96 hours. Mean scores at each timepoint are provided. The total range is 0 (no pain) to 10 (worst possible pain). Higher values on the scale represent worst outcome
Time Frame: 0-24hours, 24-48hours, 48-72hours, 72-96hours
Population: The superiority of EXPAREL admixed to bupivacaine HCI was evaluated using the Efficacy Analysis Set with the worst observation carried forward (WOCF)/interpolation method. A one-sided hypothesis test was performed at alpha=0.025 level of significance comparing EXPAREL admix and bupivacaine HCI.
  The number analyzed in one or more rows differs from overall number analyzed due to participant discontinuation in bupivacaine HCI arm and a missed assessment (protocol deviation) in EXPAREL admix arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 + 2 EXPAREL ADMIX ARM | Cohort 1 + 2 BUPIVACAINE HCI ARM
Number analyzed (Participants) | 85 | 81
units on a scale
  Worst pain at 24 hours | 8.6 (1.63) | 8.7 (1.77)
  Worst pain at 48 hours: number analyzed (Participants) | 85 | 78
  Worst pain at 48 hours | 7.9 (1.98) | 8.2 (1.81)
  Worst pain at 72 hours: number analyzed (Participants) | 84 | 78
  Worst pain at 72 hours | 6.8 (2.33) | 7.5 (2.14)
  Worst pain at 96 hours: number analyzed (Participants) | 85 | 78
  Worst pain at 96 hours | 6.6 (2.24) | 7.0 (2.34)
  Average pain at 24 hours | 6.7 (1.89) | 6.6 (2.00)
  Average pain at 48 hours: number analyzed (Participants) | 85 | 78
  Average pain at 48 hours | 5.8 (2.03) | 6.2 (1.84)
  Average pain at 72 hours: number analyzed (Participants) | 84 | 78
  Average pain at 72 hours | 5.2 (2.14) | 5.7 (2.08)
  Average pain at 96 hours: number analyzed (Participants) | 85 | 78
  Average pain at 96 hours | 4.8 (2.18) | 5.2 (1.96)
Statistical Analysis 1: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.3674, ANCOVA — Worst pain 0-24 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.1, 95% CI 2-sided [-0.6 to 0.4], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.1016, ANCOVA — Worst pain 24-48 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.4, 95% CI 2-sided [-0.9 to 0.2], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.0215, ANCOVA — Worst pain 48-72 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.7, 95% CI 2-sided [-1.4 to -0.0], Standard Error of Mean 0.34
Statistical Analysis 4: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.0794, ANCOVA — Worst pain 72-96 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.5, 95% CI 2-sided [-1.2 to 0.2], Standard Error of Mean 0.34
Statistical Analysis 5: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.3606, ANCOVA — Average pain 0-24 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.29
Statistical Analysis 6: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.0184, ANCOVA — Average pain 24-48 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.6, 95% CI 2-sided [-1.1 to -0.0], Standard Error of Mean 0.28
Statistical Analysis 7: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.0476, ANCOVA — Average pain 48-72 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.31
Statistical Analysis 8: Comparison: Cohort 1 + 2 EXPAREL ADMIX ARM vs Cohort 1 + 2 BUPIVACAINE HCI ARM; Test type: Superiority; p = 0.0529, ANCOVA — Average pain 72-96 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.31

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the date and time on or after the start date and time of study drug administration through post-operative Day 14
Description: Participants were expected to volunteer information about adverse events that they experienced. In addition, the investigator or designee questioned the patient at each scheduled time point/visit about adverse events and recorded these as well as other adverse events at the time point/visit
Arm/Group | Cohort 1 + 2 EXPAREL ADMIX ARM | Cohort 1 + 2 BUPIVACAINE HCI ARM
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/81
Serious Adverse Events (participants affected / at risk) | 3/85 | 3/81
Other Adverse Events (participants affected / at risk) | 77/85 | 71/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 + 2 EXPAREL ADMIX ARM (N=85) | Cohort 1 + 2 BUPIVACAINE HCI ARM (N=81)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 + 2 EXPAREL ADMIX ARM (N=85) | Cohort 1 + 2 BUPIVACAINE HCI ARM (N=81)
Nausea (Gastrointestinal disorders) | 34 (36) | 30 (32)
Constipation (Gastrointestinal disorders) | 30 (31) | 31 (31)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (12) | 9 (10)
Insomnia (Psychiatric disorders) | 5 (5) | 13 (14)
Headache (Nervous system disorders) | 13 (14) | 2 (3)
Hypotension (Vascular disorders) | 3 (4) | 8 (8)
Hypertension (Vascular disorders) | 5 (5) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Tachycardia (Cardiac disorders) | 4 (5) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restrictions include:

* PIs or any other party are not allowed to publish any publication for a period of twelve months following completion of the clinical study report for the trial.
* PIs or any other party shall submit a proposal to the Sponsor for approval to obtain trial results that have not been previously made public and any publication, abstract or paper or other written materials to the trial shall be submitted to the Sponsor at least 60 days prior to submission.

DOCUMENTS (2):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT05139030/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05139030/SAP_001.pdf